CLINICAL TRIAL: NCT02926872
Title: SCREENING FOR LYSOSOMAL ACID LIPASE DEFICIENCY AS THE UNDERLYING SOURCE OF HEPATIC INJURY IN PEDIATRIC PATIENTS WITH EVIDENCE OF ABNORMAL CLINICAL OR BIOCHEMICAL TESTS (DETECT)
Brief Title: Screening for Lysosomal Acid Lipase Deficiency
Status: Terminated | Type: Observational
Why Stopped: Study scope re-assessed.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-LAL-502
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: Screening; Hepatic Injury; Pediatric Patients
MeSH Terms: conditions — Wolman Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A stored (Dried Blood Spot) DBS card is collected for future assay development may be used irrespective of a patient's DBS LAL enzyme activity result.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Entire Study Population: Male or female patients who are between 2 and 16 years of age (inclusive) will be eligible for the study if they meet all components of Criterion A and/or Criterion B below, provided that these abnormalities are of unknown or unconfirmed etiology and the patient has not previously had a normal LAL enzyme activity result, has not received treatment with sebelipase alfa (Kanuma), and has no evidence of neurological dysfunction within the past year. (Note: Female patients who are of childbearing potential or are pregnant may participate in this study.)
  Interventions: Other: There is no intervention in the study

INTERVENTIONS:
Other: There is no intervention in the study

SUMMARY:
The primary outcome of this study is the development of a clinical profile of pediatric patients with LAL-D, which will enable the Sponsor to provide more focused guidance to the medical community as to which pediatric patients should be tested for LAL-D.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient is ≥ 2 to ≤ 16 years of age at the date of informed consent. (Note: Female patients who are of childbearing potential or are pregnant may participate in this study.)
2. Patient or patient's parent or legal guardian (if applicable) consents to participation in the study. If the patient is of minor age, he/she is willing to provide assent where required per local regulations, and if deemed able to do so.
3. Patient meets all components of Criterion A and/or Criterion B below.

Criterion A: Patient has dyslipidemia, defined as having at least one of the following lipid abnormalities based on a local laboratory result obtained within 3 months prior to the date of informed consent (or at the screening visit, as applicable):

LDL-c ≥ 130 mg/dL HDL c ≤ 40 mg/dL (male patients) or ≤ 50 mg/dL (female patients) Note: For patients receiving a lipid-lowering medication (LLM), the patient must have been on a stable dose of the LLM for at least 4 weeks prior to the serum lipid result.

AND

Patient has at least one of the following liver or spleen abnormalities:

Hepatomegaly, as determined by the investigator based on a physical examination or imaging procedure; Splenomegaly, as determined by the investigator based on a physical examination or imaging procedure; ALT >75 U/L or ALT >1.5x the upper limit of normal (ULN) (based on age- and gender-specific normal ranges of the local laboratory performing the assay) within 3 months prior to the date of informed consent (or at the screening visit, as applicable).

Criterion B: Patient has steatosis (microvesicular or mixed macro/microvesicular), hepatic fibrosis, and/or cirrhosis of unknown etiology, as determined from a liver biopsy performed within the previous 3 years. (Note: For patients who have received a liver transplantation, the liver biopsy results must have been obtained prior to the date of the liver transplantation.)

Exclusion Criteria:

1. Patient has a confirmed cause of liver disease other than LAL-D.
2. Patient has genetically confirmed heterozygous familial hypercholesteremia or other secondary causes of hypercholesterolemia.
3. Patient has current evidence of neurological dysfunction and/or a history of neurological dysfunction within one year prior to the date of informed consent.
4. Patient has been previously screened for LAL-D and found to have normal enzyme activity based on the reference range of the laboratory performing the assay.
5. Patient is currently receiving treatment with sebelipase alfa (Kanuma) or has previously participated in a clinical study with sebelipase alfa (Kanuma).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male or female patients who are between 2 and 16 years of age (inclusive) will be eligible for the study if they meet all components of Criterion A and/or Criterion B below, provided that these abnormalities are of unknown or unconfirmed etiology and the patient has not previously had a normal LAL enzyme activity result, has not received treatment with sebelipase alfa (Kanuma), and has no evidence of neurological dysfunction within the past year. (Note: Female patients who are of childbearing potential or are pregnant may participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Eligibility Criteria for LAL-D diagnosed patients | Confirmed LAL-D diagnosed patients, for a period extending up to a maximum of 6 months after the date of diagnosis
  Eligibility criteria will be summarized descriptively by LAL-D diagnostic status. Statistical differences in the distributions of eligibility criteria by diagnostic status will be assessed with t test for continuous variables (e.g., lab values) and chi-square test/Fishers exact test for categorical variables (e.g., presence of hepatomegaly). Among those with confirmed LAL-D, demographic data (e.g., age, sex, race/ethnicity, and country of origin) and clinical data (i.e., laboratory values, imaging and biopsy data, medications, physical exam findings, medical history, and family medical history) will be summarized as appropriate

SECONDARY OUTCOMES:
LIPA gene mutations for LAL-D diagnosed patients | Confirmed LAL-D diagnosed patients, for a period extending up to a maximum of 6 months after the date of diagnosis
  Among patients with a confirmed diagnosis of LAL-D, specific LIPA gene mutations and type of mutation will be summarized. Listings will present patient characteristics, including signs, symptoms, and laboratory values by mutation. Patient (e.g., age) and clinical features (e.g., laboratory values, signs, and symptoms) will be summarized by genetic mutation to assess associations between phenotypes and genetic variants.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No